CLINICAL TRIAL: NCT01391169
Title: Pedicled Seromuscular Flap For Enforcement Of High Risk Intestinal Anastomoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: mansoura university, mansoura university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: seromuscular flap
Record Dates: First submitted 2011-07-06; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2009-04

CONDITIONS: Peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1sup group (Active Comparator): enforcement of the anastomoses with seromuscular flap
  Interventions: Other: seromuscular flap enforcement
- 2nd group (Placebo Comparator): primary anastomosis without enforcement
  Interventions: Other: seromuscular flap enforcement

INTERVENTIONS:
Other: seromuscular flap enforcement — seromuscular flap enforcement
  Other Names: primary anastomosis only

SUMMARY:
This is a control matched prospective study evaluating the use of seromuscular flap for high risk anastomoses.

DETAILED DESCRIPTION:
30 eligible patients have been enrolled in the study then each case was matched to a control of patients who undwerwent resection anastomosis with primary anastomosis only in the same study period in terms of age, gender, comorbidity, diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* all patients with high risk anastomoses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
anastomotic leak | 5 weeks

SECONDARY OUTCOMES:
operative time | 2 hours
wound complications | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ramadan ellithy, MD, Study Director — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Mansoura, Egypt